CLINICAL TRIAL: NCT01639053
Title: U.S. Postapproval Study of Sientra Silicone Gel Breast Implants
Brief Title: Sientra Post-Approval Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tiger Biosciences, LLC. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-1007
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Breast Augmentation; Breast Reconstruction; Breast Revision
Keywords: Breast Augmentation; Breast Reconstruction; Breast Revision; Silicone breast implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gel Participants
- Control Participants

SUMMARY:
This is a ten-year postapproval study to evaluate the long-term clinical performance of Sientra Silicone Gel Breast Implants under general conditions of use in the postmarket environment.

ELIGIBILITY:
Inclusion Criteria:

1. Genetic female with US residency
2. Is at least 18 years old for primary or revision reconstruction or 22 years old for primary or revision augmentation
3. Agrees to Sientra study requirements

Exclusion Criteria:

1. Has an active infection anywhere in body
2. Has active cancer without adequate treatment
3. Currently pregnant or nursing
4. Has any condition or diagnosis that, in the investigator's opinion, would negatively affect ability to complete study requirements
5. If control participant, has undergone breast implant surgery with silicone gel-filled breast implants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who receive Sientra Silicone Gel Breast Implants for augmentation, revision augmentation, reconstruction, and revision reconstruction. Control participants are candidates for and undergo aesthetic surgery other than implantation with Silicone Gel Breast implants.
Sampling Method: Non-Probability Sample
Enrollment: 5498 (Actual)
Dates: Start 2012-04; Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Long-term safety of Sientra Silicone Gel Breast Implants in women | 10-years

CONTACTS AND LOCATIONS:
Overall Officials: Sientra, Inc., Study Director — Sponsor GmbH
Locations (1):
- Sientra, Inc., Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No